CLINICAL TRIAL: NCT05514249
Title: Treatment of a Single Patient With CRD-TMH-001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cure Rare Disease, Inc (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-CRD-TMH-001
Record Dates: First submitted 2022-08-11; First posted 2022-08-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; Muscular Dystrophy; CRISPR; gene-editing
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Masking Description: Single patient clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single patient (Experimental): Single dose of CRD-TMH-001 administered by IV
  Interventions: Drug: CRD-TMH-001

INTERVENTIONS:
Drug: CRD-TMH-001 — Participant will receive a single dose of CRD-TMH-001 administered via intravenous injection.

SUMMARY:
The study is a single patient study intended to understand the effects of a gene-editing therapeutic to treat a rare mutation of Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
The objective of the study is to assess the safety and preliminary efficacy of CRD-TMH-001 after intravenous administration for a period of 1 year with long-term follow-up out to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Completion of informed consent
* Confirmation of genetic mutation
* Confirmation of absence of elevated AAV9 NAbs

Exclusion Criteria:

- Any significant medical issue(s) (past or current) that would, in the opinion of the Principal Investigator (PI), prevent this patient from being dosed.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of CRD-TMH-001 | 1 year
  To assess the safety and tolerability of the therapeutic by measuring both serious and non-serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Wong, MD, Principal Investigator — UMass Chan Medical School; Medical Affairs, Study Director — Cure Rare Disease
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No